CLINICAL TRIAL: NCT00202631
Title: Abdominal Functional Electrical Stimulation to Augment Breathing in Tetraplegia
Brief Title: Abdominal Functional Electrical Stimulation in Tetraplegia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: South Glasgow University Hospitals NHS Trust (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AbdomGlasgow
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2006-11-28 (Estimated); Status verified 2006-11

CONDITIONS: Tetraplegia; Spinal Cord Injury
Keywords: tetraplegia; quadriplegia; spinal cord injury; functional electrical stimulation; abdominal stimulation
MeSH Terms: conditions — Quadriplegia; Spinal Cord Injuries

INTERVENTIONS:
Device: Surface Functional Electrical Stimulation

SUMMARY:
People with high spinal lesions are at risk of respiratory complications because they have partial or complete paralysis of breathing muscles. Previous work has shown that tetraplegic lung volumes can be increased by using abdominal FES during expiration. The technique is attractive because it is non-invasive, painless in tetraplegia and completely reversible. It may provide a treatment for augmenting the patient's breathing both in the acute presentation of spinal injury (when half of cervical injuries require ventilation) and in long term management of tetraplegia and high paraplegia. We propose a pilot study in a small group of subjects to see if the technique is feasible from both a clinical and engineering viewpoint. The aims of the study are: 1)To examine the effects of abdominal FES on lung mechanics and gas exchange in tetraplegic subjects. 2)To optimise the stimulation pattern and intensity via electronic stimulators and to design a trigger to allow the FES to follow the subject's own breathing cycle automatically.

DETAILED DESCRIPTION:
Patients with high spinal cord injury (SCI) usually have paralysed intercostal muscles and rely on diaphragm function alone for respiration. They have low tidal volumes and inadequate cough. These patients are vulnerable to respiratory complications in the immediate post-injury phase and remain at life-long risk of chest problems. Usual treatments include intensive physiotherapy and intermittent positive pressure ventilation to augment the patient's tidal volume and to help clear excess secretions.

Tidal volumes can also be increased by electrical stimulation of the surface of abdominal muscles during expiration. During stimulation the patient expires below functional residual capacity (the amount of air left after normal expiration). The natural elasticity of the chest wall then causes a recoil increase in the size of the next inspired breath. Functional electrical stimulation (FES) of the abdominal muscles is theoretically an attractive technique to augment respiration. It is non-invasive, it mimics natural physiological processes and tetraplegic patients cannot sense abdominal discomfort. There are potential applications in acute SCI patients to prevent the need for artificial ventilation and to aid ventilator weaning. The technique could also be used in chronically injured patients to augment ventilation.

Clinical staff at the Queen Elizabeth National Spinal Injuries Unit have collaborated extensively with engineering and bioengineering teams from Glasgow University and the University of Strathclyde in the use of FES in SCI. FES is already being used successfully in the Unit for paraplegic cycling and upper limb exercise in tetraplegia. We have performed abdominal FES on one SCI subject with complete diaphragm paralysis and produced a tidal volume of one hundred millilitres (McLean and Hunt, unpublished observation).

Before starting a large scale project it is important to confirm whether we can reliably reproduce at least some of the findings of Stanic et al. It would be very interesting if we could show any change in gas exchange as well as simply increasing tidal volume. Engineering issues include optimisation and programming of the FES stimulus. We propose a pilot study in QENSIU to establish whether the technique is of practical benefit to spinal cord injured patients.

ELIGIBILITY:
Inclusion Criteria:

* cervical spinal cord injury

Exclusion Criteria:

* subject must not be ventilator-dependent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 4
Dates: Start 2002-06; Study Completion 2006-11

PRIMARY OUTCOMES:
Tidal Volume
Peak Expiratory Flow

SECONDARY OUTCOMES:
Expired CO2 levels
Vital Capacity

CONTACTS AND LOCATIONS:
Overall Officials: Alan N McLean, MRCP, Principal Investigator — Queen Elizabeth National Spinal Injuries Unit, Glasgow; Kenneth J Hunt, BSc, PhD, DSc, Principal Investigator — Department of Mechanical Engineering, University of Glasgow
Locations (1):
- Queen Elizabeth National Spinal Injuries Unit, Glasgow, Lanarkshire, United Kingdom

REFERENCES:
- [Background] Stanic U, Kandare F, Jaeger R, Sorli J. Functional electrical stimulation of abdominal muscles to augment tidal volume in spinal cord injury. IEEE Trans Rehabil Eng. 2000 Mar;8(1):30-4. doi: 10.1109/86.830946. PMID 10779105